CLINICAL TRIAL: NCT05415046
Title: Retrospective Analyses of Sacral Erector Spinae Plane Blocks in Pediatric Patients: Is it Time to Discuss the Necessity of Caudal Block
Brief Title: Sacral Erector Spinae Plane Blocks in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Can AKSU, MD, Principal investigator., Kocaeli University
Other Study IDs: GOKAEK-2021/6.04
Record Dates: First submitted 2022-06-04; First posted 2022-06-10 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sacral ESPB: Sacral erector spinae plane block performed with 0,25% bupivacaine (1 mL/kg-max 20mL), under general anesthesia before the start of the surgery.
  Interventions: Procedure: Sacral ESPB

INTERVENTIONS:
Procedure: Sacral ESPB — Erector spinae plane block performed with 0,25% bupivacaine (1 mL/kg-max 20mL), under general anesthesia before the start of the surgery.

SUMMARY:
Patients who were operated by Department of Pediatric Surgery and who received sacral erector spinae plane blocks as a part of postoperative analgesia management will be scanned.

DETAILED DESCRIPTION:
Erector spinae plane block (ESPB) is a safe and effective regional anesthesia technique in pediatric patients and can be performed at any level of the thoracic and lumbar vertebrae. In addition, ESPB can be performed at the sacral region in the midline. In pediatric patients, sacral ESPB provides effective analgesia and this method can replace caudal blocks.

This study aims to investigate the efficacy of sacral ESPB retrospectively. Demographical data of the patient, indication/surgery type, total volume applied, additional analgesic use, type of the analgesic if used will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were operated by Department of Pediatric Surgery

Exclusion Criteria:

* Incomplete patient forms

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients who were operated by Department of Pediatric Surgery and performed sacral ESPB for postoperative analgesia.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Face, Legs, Activity, Cry, Consolability (FLACC) Scale | Postoperative 24th hour.
  The scale is scored in a range of 0-10 with 0 representing no pain (meaning a better outcome). The scale has five criteria, which are each assigned a score of 0, 1 or 2.
Rescue analgesic-paracetamol | During the postoperative 24th hour.
  The need and amount of the IV paracetamol given
Rescue analgesic-ibuprofen | During the postoperative 24th hour.
  The need and amount of the oral ibuprofen given

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No